CLINICAL TRIAL: NCT03875716
Title: A Phase 2 Study of De-Intensified Risk-Adapted Postoperative Radiation Therapy for Human Papilloma Virus Associated Oropharyngeal Squamous Cell Carcinoma: the ADAPT Trial
Brief Title: Study of De_Intensified Postoperative Radiation Therapy for HPV Associated Oropharyngeal Squamous Cell Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Danielle Margalit, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-009
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Low Risk (Experimental): Observation without adjuvant therapy
  * Pathologic T0-2, N0-1
  * Minimum of 15 lymph nodes retrieved on neck dissection per dissected side of the neck
  * Single positive lymph node up to 3cm
  * No extranodal extension
  * Clear margins
  * Undetectable postoperative circulating tumor HPV DNA
  Interventions: Radiation: Radiation therapy
- Intermediate Risk (Experimental): Reduced-dose radiation (46Gy)
  * Pathologic T0-2N0-2 and any one of the following features:
  * 2 or more positive lymph nodes
  * single node >3cm
  * <15 lymph nodes retrieved on neck dissection for each side of the neck
  * Positive lymph nodes in level IB, IV, or V
    -≤1mm extranodal extension
  * Positive lymph node(s) contralateral to the primary tumor
  * Close margins
  * Detectable postoperative circulating tumor HPV DNA
  Interventions: Radiation: Radiation therapy
- High Risk (Experimental): Postoperative radiation (60Gy) without chemotherapy
  * Pathologic T0-4N0-2 and any one of the following features:
    ->1mm extranodal extension
  * Microscopic positive margins
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — Radiation therapy

SUMMARY:
This research study is studying lowering the standard dose of radiation and chemotherapy after surgery, to minimize the side effects and improve the quality of life.

DETAILED DESCRIPTION:
This research study is being done to study if less intensive treatments can be used after surgery for head and neck cancers that are due to the human papilloma virus (HPV). In general, these cancers have better cure rates than other types of head and neck cancers. Therefore, the investigators are studying whether we can safely reduce the amount of treatment after surgery, such as surveillance (instead of using radiation) or less radiation or less chemotherapy, while maintaining good cure rates. The investigators hope that by reducing the intensity of treatment, this will lead to less side effects during and after cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous cell carcinoma of the tonsil or base of tongue (oropharynx) or unknown primary with p16-positive cervical lymph node metastases
* HPV-associated tumor as defined by: positive p16 immunohistochemistry (>70%) OR in situ hybridization OR PCR-based methods
* Eligible for curative-intent surgery with anticipated negative margins
* Surgery performed at Brigham & Women's Hospital
* Age 18 or older years.
* ECOG performance status 0-1 (Karnofsky ≥70%, see Appendix A)
* Normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,000/mcL
  * platelets ≥100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine ≤ 1.5 times the institutional upper limit of normal OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* Patients with ≤20 pack-years of cumulative cigarette smoking. Pack-years are calculated by multiplying the number of years smoked with the pack of cigarettes smoked per day. One pack is considered to contain 20 cigarettes.
* Tumor clinical stage (AJCC 8th edition): T0 or T1 or T2
* Nodal clinical stage (AJCC 8th edition): N0 or N1
* No distant metastases. Clinical M-stage must be M0 (AJCC 8th edition).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior history of head and neck cancer within 5 years.
* Prior head and neck radiation
* Clinically fixed or matted nodes
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Note: that HIV positive patients will be eligible.
* Pregnant women are excluded from this study because of the teratogenic risks of radiation exposure to the developing fetus. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with radiation therapy and supportive care medications required for symptomatic management of head and neck cancer side effects as well as general anesthesia required for oncologic head and neck surgery, breastfeeding should be discontinued if the mother is enrolled in the study. Pregnancy status will be determined by a serum pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 2 years
  Survival without any signs or symptoms of cancer after the treatment ends.

SECONDARY OUTCOMES:
Overall Survival | 2 years
  The length of time from the start of treatment until death.
Toxicity Rate | 2 years
  Adverse events experienced by the participants.
Quality Of Life Questionnaire | 2 Years
  Assesses the physical; social/family; emotional and functional wellbeing, using Functional Assessment of Cancer Therapy for Head and Neck (FACT-H&N) on a scale of 0-4 (where 0 indicates the lowest quality of life and 4 indicates the highest quality of life).
Symptom burden: | 2 years
  Patient-reported symptom severity, using M.D. Anderson Symptom Inventory - Head & Neck (MDASI-HN) on a scale of 0-10 (where 0 indicates symptom is not present and 10 indicates the symptom is as bad as can be)
Dysphagia | 2 Years
  Swallowing ability or difficulty. Dysphagia-related quality of life, assessed with the MD Anderson Dysphagia Inventory (MDADI) on a scale of 1-5 (where 1 indicates the patient strongly agrees and 5 indicates the patient strongly disagrees)
Shoulder dysfunction | 2 Years
  Shoulder function or dysfunction is measured with the "neck dissection impairment index" (NDII). This evaluates how much the patient's neck and/or shoulder affects them as a result of the treatment they received in their neck during the overall management of their cancer. This scale goes from 1-5 (1 being "not at all" and 5 being "a lot")

CONTACTS AND LOCATIONS:
Overall Officials: Danielle N. Margalit, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation